CLINICAL TRIAL: NCT07374276
Title: Brain-Computer Interface (BCI) With Virtual Reality (VR) in Upper Limb Rehabilitation After Stroke: A Randomized Crossover Clinical Trial
Brief Title: BCI With Virtual Reality for Stroke Rehabilitation: A Crossover Study
Acronym: NOISyS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Lisbon (Other)
Collaborators: Centro de Medicina de Reabilitação de Alcoitão (Unknown)
Responsible Party: Principal Investigator, Athanasios Vourvopoulos, Principal Investigator, Technical University of Lisbon
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1801P.01287; 10.54499/2022.02283.PTDC (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia (FCT))
Record Dates: First submitted 2025-12-09; First posted 2026-01-28 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: Stroke; Brain-Computer Interface; Virtual Reality; Motor Imagery; Upper Extremity; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Each participant will complete two intervention periods, corresponding to two different intervention types (MI-VR-BCI or MI-BCI), administered in a randomized order. A 3-week washout period will separate the two intervention periods. Pre- and post-intervention assessments will be conducted for each period, resulting in a total of four assessments per participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI-VR-BCI Training (Experimental): Participants will perform motor imagery-based brain-computer interface training combined with immersive virtual reality and multimodal feedback (visual, auditory, and haptic).
  Interventions: Device: Motor Imagery-based Brain-Computer Interface coupled with Virtual Reality (MI-BCI-VR)
- MI-BCI (Active Comparator): Participants will perform motor imagery-based brain-computer interface (MI-BCI) training based on a cue-based protocol.
  Interventions: Device: Motor Imagery-based Brain-Computer Interface (MI-BCI)

INTERVENTIONS:
Device: Motor Imagery-based Brain-Computer Interface coupled with Virtual Reality (MI-BCI-VR) — The training paradigm will involve motor imagery coupled with EEG-based BCI control and immersive virtual reality (VR) feedback. VR feedback will consist of NeuRow, a first-person perspective training paradigm that allows multimodal visual, auditory and haptic feedback through the use of immersive virtual reality headset and haptic controllers. Sessions will have a frequency of 3 times per week, during 6 weeks.
  Arms: MI-VR-BCI Training
Device: Motor Imagery-based Brain-Computer Interface (MI-BCI) — The training paradigm will involve motor imagery combined with EEG-based BCI control using a cue-based visual paradigm. Sessions will be conducted three times per week over a period of six weeks.
  Arms: MI-BCI

SUMMARY:
The goal of this clinical trial is to investigate if training sessions of motor imagery associated with brain-computer interface and motor observation through virtual reality (MI-VR-BCI) can help to improve arm and hand recovery after a stroke. The main questions to answer are:

* Can adding MI-BCI-VR sessions improve upper limb movement?
* Can it help stroke survivors perform daily activities more easily?
* Does this type of training improve brain activity and connections related to movement?

Researchers will compare this type of intervention with motor imagery associated with a standard brain-computer interface intervention (MI-BCI) to see if there are added effects to upper limb function, activity and brain connections.

Participants will :

* Perform two intervention periods in a random order: one with MI-VR-BCI training sessions and other with MI-BCI training sessions. Each period will involve 3 weekly sessions of training, during 6 weeks, with the intervention periods being separated by 3 weeks.
* Complete four assessment sessions: one at the beginning and another at the end of each intervention period.

DETAILED DESCRIPTION:
Stroke is a leading cause of long-term disability worldwide, often resulting in upper limb (UL) impairment. Approximately 70% of stroke survivors experience UL dysfunction, with a significant portion continuing to show deficits into the chronic phase. This impacts independence and quality of life, highlighting the need for effective rehabilitation strategies.

Brain-Computer Interface (BCI) interventions have shown promise in improving UL function by enabling patients to modulate brain activity through neurofeedback in a closed-loop system. When combined with multisensory feedback (visual, auditory, and somatosensory) BCIs may promote neuroplasticity and motor recovery. The use of Motor Imagery (MI) and embodied Virtual Reality (VR) may further enhance motor learning by reinforcing motor patterns and creating meaningful, immersive rehabilitation experiences.

Despite encouraging evidence, the clinical and neurophysiological benefits of combining BCI with VR and MI remain underexplored, particularly when associated with longer intervention periods, the impact in activities of daily living and the influence of patient-specific traits such as motor, cognitive, or behavioral dimensions. In light of these considerations, the primary objectives of this study are:

* To assess the preliminary effects of applying a motor imagery based Brain-Computer Interface with Virtual Reality (MI-BCI-VR) paradigm on upper limb function and activity in individuals with stroke.
* To evaluate the neurophysiological effects of this intervention on brain activity and its relationship with clinical measures of upper limb function.

The secondary objectives of the study are:

* To explore the influence of individual characteristics on clinical outcomes and neurophysiological changes observed.
* To examine the specific contribution of embodied Virtual Reality associated with BCI in upper limb rehabilitation after stroke.
* To understand participant's experience with the different intervention paradigms, including acceptability and usability, and to inform the technology development process.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stroke confirmed by neuroimaging, with resulting upper limb hemiparesis.
* Time since stroke between 6 and 24 months at the time of selection.
* Sufficient cognitive ability to understand and follow the intervention procedures.
* Spasticity score <3 on the Modified Ashworth Scale in upper limb muscle groups.
* Adults aged 18 to 80 years.
* Ability to remain seated for approximately 2 hours.
* Motivation to participate and capacity to provide informed consent.
* Undergoing conventional rehabilitation therapy during the study period.

Exclusion Criteria:

* Severe communication difficulties preventing comprehension or execution of instructions.
* Skin lesions, allergies, or metal implants in the cephalic region, or history of craniectomy, that hinder electrode placement or interfere with EEG signal acquisition.
* Concomitant neurological or musculoskeletal conditions affecting upper limb motor function.
* Other neurological, musculoskeletal, or psychiatric conditions that may compromise participation or study outcomes (e.g., major depression, severe visual impairment, photosensitive epilepsy, frequent vertigo or dizziness).
* Upper limb impairment due to a previous stroke.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in Upper Limb Motor Function (Fugl-Meyer Assessment - Upper Extremity) | Baseline and end of each 6-week intervention period (up to 15 weeks total, including washout).
  Within-subject difference in the change in upper limb motor function, as assessed by the Fugl-Meyer Assessment for the Upper Extremity (FMA-UE), between the two intervention conditions (MI-BCI-VR vs. MI-BCI). FMA-UE scores range from 0 to 66, with higher scores indicating better motor function and less impairment.
Change in Upper Limb Activity (Action Research Arm Test - ARAT) | Baseline and end of each 6-week intervention period (up to 15 weeks total, including washout).
  Within-subject difference in the change in upper limb activity, as assessed by the Action Research Arm Test (ARAT), between the two intervention conditions (MI-BCI-VR vs. MI-BCI). The ARAT is a standardized measure that evaluates upper limb functioning through tasks involving grasp, grip, pinch, and gross movement. Scores range from 0 to 57, with higher scores indicating better functional ability. This outcome assesses the impact of the intervention on functional use of the affected arm in daily activities.
Change in EEG Event-Related Desynchronization/Synchronization (ERD/ERS) | During each intervention session across both 6-week intervention periods (up to 15 weeks total, including washout).
  Changes in event-related desynchronization and synchronization (ERD/ERS) during motor imagery tasks, derived from EEG recordings to assess intervention-related modulation of sensorimotor cortical activity.
Change in EEG Hemispheric Lateralization Index | During each intervention session across both 6-week intervention periods (up to 15 weeks total, including washout).
  Changes in EEG-derived hemispheric lateralization indices during motor imagery tasks, used to evaluate intervention-related reorganization of cortical motor networks.
Change in EEG Connectivity Measures | During each intervention session across both 6-week intervention periods (up to 15 weeks total, including washout).
  Exploratory changes in EEG-based functional connectivity metrics between motor-related cortical regions during motor imagery tasks.

OTHER OUTCOMES:
Cognitive Function (Montreal Cognitive Assessment - MoCA) | Baseline and end of each 6-week intervention period (up to 15 weeks total, including washout).
  Cognitive function will be assessed using the MoCA to characterize participants' baseline function, explore potential changes associated with the intervention, and examine its role as a predictor or moderator of rehabilitation outcomes. The MoCA is a brief cognitive screening tool designed to assess multiple cognitive domains with a score ranging from 0 to 30, with higher scores reflecting better cognitive performance.
Stroke Patient Participation (Stroke Impact Scale - SIS) | Baseline and end of each 6-week intervention period (up to 15 weeks total, including washout).
  Stroke-related participation and quality of life, as measured by the SIS 2.0, will be used to characterize participants' baseline function, explore potential changes associated with the intervention, and examine its role as a predictor or moderator of rehabilitation outcomes. The SIS is a self-report questionnaire designed to assess the impact of stroke across multiple domains, including strength, hand function, mobility, communication, memory, emotion, activities of daily living (ADL), and social participation. Higher scores indicate better perceived recovery and participation.
Depressive Symptoms (Patient Health Questionnaire-9 - PHQ-9) | Baseline and end of each 6-week intervention period (up to 15 weeks total, including washout).
  Depressive symptoms will be assessed using the PHQ-9 to characterize participants' baseline function and explore their potential role as a predictor or moderator of rehabilitation outcomes. PHQ-9 is a self-report questionnaire with 9 items used to screen for and measure the severity of depressive symptoms. Each item is rated on a 4-point scale (0-3), with higher total scores indicating greater depressive symptomatology.
Spatial Neglect (Bells Test) | Baseline and end of each 6-week intervention period (up to 15 weeks total, including washout).
  Spatial Neglect will be screened using the Bells Test to characterize participants' baseline function, explore potential changes associated with the intervention, and examine its role as a predictor or moderator of rehabilitation outcomes. The Bells Test is a paper-and-pencil cancellation task allowing the evaluation of egocentric neglect in peripersonal space through the analysis of the number and spatial distribution of omissions
Upper Limb Spasticity (Modified Ashworth Scale - MAS) | Baseline and end of each 6-week intervention period (up to 15 weeks total, including washout).
  Spasticity in the upper limb will be assessed using the MAS to describe muscle tone at baseline, to explore potential changes associated with the intervention, and examine its role as a predictor or moderator of rehabilitation outcomes. The MAS is a 6-point ordinal scale ranging from 0 to 4, with higher scores indicating greater spasticity levels.
Intervention and Technology Assessment (Questionnaire) | Immediately after completion of each 6-week intervention period (2 assessment points per participant).
  Participants' experience with the intervention and interaction with the technology will be quantitatively assessed using a questionnaire developed by the research team, covering multiple dimensions (setup, session experience, visual scenario and interaction, task execution, gamification and feedback, and potential adverse effects). The instrument includes 5-point Likert scale items and visual analogue scale components.
Participant Experience and Acceptability of the Intervention (Qualitative Assessment) | After completion of both intervention periods (end of study).
  Participants' subjective experiences, perceived usability, clinical relevance, challenges, preferences, and suggestions regarding the intervention paradigms will be qualitatively explored, through a semi-structured interview. Data will be analyzed using reflexive thematic analysis to identify recurring themes and insights.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Medicina de Reabilitação de Alcoitão, Alcabideche, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared outside the study team.

REFERENCES:
- See also: NOISyS project webpage providing an overview of the project, including objectives, consortium members, and outputs. — https://www.noisys-project.eu/